CLINICAL TRIAL: NCT01583582
Title: Assessment on Antihypertensive Effect and Safety of Bioactive Peptides Derived From Coldwater Shrimp (Pandalus Borealis) in Healthy Subjects With Mild or Moderate Hypertension
Brief Title: Antihypertensive Effect and Safety of Peptides Derived From Coldwater Shrimp
Acronym: MARE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marealis AS (Industry)
Responsible Party: Principal Investigator, Niina Tapola, Project Manager, Marealis AS
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MARE-050312
Record Dates: First submitted 2012-04-20; First posted 2012-04-24 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Hypertension; Blood Pressure
Keywords: randomized double-blind placebo-controlled study; peptide concentrate; Coldwater Shrimp; antihypertensive effect; mild hypertension; moderate hypertension; blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Refined peptide concentrate, 1200 mg (Experimental): Refined peptide concentrate, 1 200 mg, once a day
  Interventions: Dietary Supplement: Marealis Refined Peptide Concentrate
- Refined peptide concentrate, 2 x 600 mg (Experimental): Refined peptide concentrate, 600 mg, twice a day
  Interventions: Dietary Supplement: Marealis Refined Peptide Concentrate
- Refined peptide concentrate, 0 mg (Placebo Comparator)
  Interventions: Dietary Supplement: Marealis Refined Peptide Concentrate

INTERVENTIONS:
Dietary Supplement: Marealis Refined Peptide Concentrate — 1200 mg per os, once a day, 8 weeks
  Arms: Refined peptide concentrate, 1200 mg
Dietary Supplement: Marealis Refined Peptide Concentrate — 600 mg per os, twice a day, 8 weeks
  Arms: Refined peptide concentrate, 2 x 600 mg
Dietary Supplement: Marealis Refined Peptide Concentrate — 0 mg per os, daily, 8 weeks
  Arms: Refined peptide concentrate, 0 mg

SUMMARY:
The purpose of this proof of concept study is to find out the efficacy of Marealis Refined Peptide Concentrate (RPC) from Coldwater Shrimp (Pandalus borealis) containing ACE-inhibiting peptides on blood pressure in subjects with mild or moderate hypertension.

ELIGIBILITY:
Inclusion Criteria:

* mild or moderate hypertension (systolic blood pressure 130 - 160 mmHg and diastolic blood pressure ≤ 100 mmHg)
* age 30 - 75 years
* body weight ≥ 60 kg
* stable body weight
* use of effective contraception in women of childbearing potential

Exclusion Criteria:

* body mass index ≥ 35
* antihypertensive drug treatment, regular high dose NSAID treatment and the use of cyclosporine or tacrolimus
* diabetes (type 1 and 2)
* anemia, abnormal electrolytes, proteinuria, abnormal liver, kidney and thyroid function, clinically significant biochemistry, any other clinically significant hematology and/or biochemistry at the investigator's discretion
* cardiovascular disease (myocardial infarction, unstable angina pectoris, coronary artery bypass graft, percutaneous transluminal coronary angioplasty, temporal ischemic attack within six months prior to screening) including stroke and congestive heart failure
* secondary hypertension history of cancer or malignant disease within the past five years
* any metabolic disease, gastrointestinal disorder or other clinically significant disease/disorder which in the investigator's opinion could interfere with the results of the study or the safety of the subjects
* fish and other seafood allergies, citrus allergy, multiple food allergies
* alcohol abuse
* smokers and tobacco/snuff/nicotine users
* consumption of food supplements targeted to blood pressure lowering within 30 days before randomization
* pregnant and lactating mothers, women, planning for pregnancy during the study
* participation in clinical trials 30 days prior to this study and participation in other clinical intervention

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
change in systolic blood pressure | from baseline after 8 weeks of treatment
  change from baseline after 8 weeks of treatment in systolic office blood pressure

SECONDARY OUTCOMES:
change in diastolic blood pressure | from baseline after 8 weeks of treatment
  change from baseline after 8 weeks of treatment in diastolic blood pressure
mean systolic blood pressure | at the end of a 8-week treatment
mean diastolic blood pressure | at the end of a 8-week treatment
change in systolic blood pressure | from baseline after 4 weeks treatment
diastolic blood pressure | from baseline after 4 weeks treatment
diastolic blood pressure | from baseline after 2 weeks treatment
mean heart rate | at the end of a 8-week treatment
mean fasting plasma glucose concentration | at the end of a 8-week treatment
mean fasting plasma lipids concentration | at the end of a 8 week treatment
  plasma total cholesterol, HDL-cholesterol, LDL-cholesterol and total triglycerides concentration, respectively
mean serum C-reactive protein | at the end of a 8-week treatment
blood count | at the end of a 8-week treatment
plasma glutamyltransferase | at the end of a 8-week treatment
plasma creatinine | at the end of a 8-week treatment
plasma sodium concentration | at the end of a 8-week treatment
plasma potassium concentration | at the end of a 8-week treatment
adverse events | during the 8-week treatment
change in systolic blood pressure | from the baseline after 2 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Essi S Sarkkinen, Ph.D, Study Director — Oy Foodfiles Ltd; Sakari A Nieminen, MD, Principal Investigator — Oy Foodfiles Ltd
Locations (1):
- Oy Foodfiles Ltd, Kuopio, Finland